CLINICAL TRIAL: NCT06721598
Title: An Open-label, Non-interventional, Single-group Follow-up Study to Evaluate the Safety and Efficacy of an Anti-CD19 CAR-T Product in Adult Patients with Relapsed or Refractory Forms of B-cell Lymphoproliferative Disorders
Brief Title: An Extension Study to Evaluate the Safety and Efficacy of an Anti-CD19 CAR-T Product in Patients with B-cell Lymphoproliferative Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Other Study IDs: HemC101-01-02
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Non-Hodgkin Lymphoma, B-cell; Acute Lymphoblastic Leukemia ALL
Keywords: CAR-T; B-cell lymphoma; non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hem101 Arm: Subjects received Hem101 in Study Hem101-01-01 will be followed for 11 month

SUMMARY:
This follow-up study is designed to evaluate the long-term safety and effectiveness of a treatment called anti-CD19 CAR-T cell therapy in adults with certain B-cell blood cancers. These cancers include types that have returned after treatment or have not responded to other therapies. CAR-T cell therapy involves using a patient's own immune cells, which are modified in a lab to specifically target and destroy cancer cells with a marker called CD19. The study will look at how well patients tolerate this treatment over time, as well as its ability to keep cancer in remission or reduce its severity.

Patients who have previously received CAR-T therapy in an earlier clinical trial and meet specific criteria can participate in this study. The research will include regular follow-up visits over approximately 11 months to monitor for side effects, assess cancer response, and track the activity of CAR-T cells in the body. This study does not involve additional treatments but focuses on understanding the long-term outcomes of CAR-T therapy to provide better care for patients in the future.

DETAILED DESCRIPTION:
This is a Phase I/II open-label, non-interventional, single-arm follow-up study evaluating the long-term safety and efficacy of anti-CD19 CAR-T cell therapy in adult patients with relapsed or refractory B-cell lymphoproliferative disorders. CAR-T cell therapy is an advanced immunotherapy that modifies a patient's T cells to target the CD19 antigen on B cells. This follow-up study focuses on assessing the durability of treatment responses and monitoring potential late-onset adverse events in patients who previously received anti-CD19 CAR-T cells during the HemC101-01-01 trial (NCT06705530).

The primary objective of this study is to evaluate the long-term safety profile of second-generation anti-CD19 CAR-T cells, including the incidence, duration, and severity of adverse events. Secondary objectives include assessing the durability of clinical responses, such as overall response rate (ORR), progression-free survival (PFS), duration of response (DoR), and overall survival (OS). Additionally, the study aims to monitor the persistence and expansion of CAR-T cells in peripheral blood and detect the development of anti-drug antibodies (ADAs) that may impact therapeutic efficacy.

Eligible participants include adults aged 18-70 who completed the HemC101-01-01 trial and meet all inclusion criteria, such as sufficient organ function and negative pregnancy tests where applicable. This study involves periodic follow-up visits over 11 months post-CAR-T cell infusion, during which clinical assessments, laboratory evaluations, and safety monitoring will be conducted. No additional CAR-T cell infusions will be administered in this follow-up study.

The trial is conducted at a single clinical center in Russia under the sponsorship of the National Medical Research Center of Hematology, Ministry of Health of Russia. The data collected will provide insights into the long-term safety and efficacy of anti-CD19 CAR-T therapy, contributing to the development of treatment protocols and improving outcomes for patients with relapsed or refractory B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Successful completion of the HemC101-01-01 study procedures.
2. Negative pregnancy test for women of reproductive potential.

Exclusion Criteria:

1. Uncontrolled life-threatening infection. A urinary tract infection is acceptable. Patients who received intravenous antibiotics before IMP administration or in whom intravenous antibiotics have not been discontinued 7 days before inclusion in the study. Prophylactic use of antibiotics, antiviral, or antifungal drugs is allowed.
2. The use of therapeutic interventions prohibited by the protocol (glucocorticosteroids, allogeneic cell therapy, GVHD therapy, chemotherapy, alemtuzumab, clofarabine, cladribine, and biologics derived from mouse materials).
3. Non-adherence to HemC101-01-01 study procedures that, in the investigator's opinion, put the patient at risk if they participate in the study and may significantly bias the assessment of study results.
4. Any clinically relevant data that, in the investigator's opinion, affects the patient's ability to enter the study and puts the patient at risk.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received the IMP in the HemC101-01-01 study and completed it per protocol
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of Treatment-Emergent Adverse Events [Safety] | 11 month starting on the 29th day after IMP administration
  Frequency of any adverse events (AEs) reported during the study period and AE characterization (severity, seriousness, etc.)
ORR [Efficacy] | 11 month starting on the 29th day after IMP administration
  Overall response rate (ORR) defined as the proportion of subjects with complete response (CR) or partial response (PR)

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Offical approval of the trial by the Ministry of Health of the Russian Federation — https://grls.rosminzdrav.ru/CIPermissionMini.aspx?CIStatementGUID=bd05c1b9-1bba-447b-aeba-9a706c387223&CIPermGUID=90f14d17-beb1-4233-8f4b-fdae1356363f